CLINICAL TRIAL: NCT00200655
Title: Safety and Efficacy of Pravastatin in Relapsing-remitting MS: a Double Blind Placebo Controlled Study
Brief Title: Safety and Efficacy of Pravastatin in Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRD/03/10-I-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2008-06

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pravastatin
Drug: Placebo

SUMMARY:
Therapeutic strategies for multiple sclerosis (MS) are essentially based on the use of immunomodulatory agents such as interferon b and glatirmere acetate, but their efficacy is quite limited, they are not well tolerated and they have a very high cost. Recent works showed an immunomodulatory effects of HMG-CoA reductase inhibitors (the so-called "statins"). In experimental allergic encephalopathy, a murine model of MS, statins inhibit the onset and progression of the disease through a shift from Th1 towards Th2 cytokine production. Other in vitro studies suggest the ability of statins to inhibit the lymphocyte migration through the blood brain barrier. Furthermore, in an open labeled human study in MS, statin regimen was associated with a decreased lesional activity assessed by MRI. Statins are well tolerated drugs, used for many years, with a low cost and with a putative efficacy in MS. The investigators suggest to test the pravastatin safety and efficacy on MRI criteria in a double-blind, placebo-controlled study in 40 patients with a relapsing-remitting MS.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting MS with diagnosis defined by the McDonald criteria (McDonald et al., 2001) with no current disease modifying therapy (interferon, copaxone or immunosuppressant drugs) since at least 3 months and an EDSS score < 5.
* At least one gadolinium positive lesion on the MRI of the selection phase is needed.
* No current statin therapy.
* Normal renal and hepatic biological tests.
* No current pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-12; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Number of gadolinium positive lesions at month 6 in each group. | at month 6 in each group

SECONDARY OUTCOMES:
Cumulated number of gadolinium positive lesions in each group after 6 months of follow-up | after 6 months of follow-up
Number of new T2 lesions

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DAMIER, MD, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France